CLINICAL TRIAL: NCT04877392
Title: Analgesic Effect of Inhaled Lavender Essential Oil for Frenotomy in Healthy Neonates: a Randomized Clinical Trial
Brief Title: Analgesic Effect of Inhaled Lavender Essential Oil for Clipping of Tongue-ties
Acronym: LEO-SME1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020/9373/I
Record Dates: First submitted 2021-04-27; First posted 2021-05-07 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2021-04

CONDITIONS: Ankyloglossia
Keywords: ankyloglossia; tongue-tie; aromatherapy; lavender; pain; neonate
MeSH Terms: conditions — Ankyloglossia; Pain | interventions — lavender oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (usual measures to control pain) (No Intervention): The neonate was taken to the neonatal unit and monitored with a pulse-oximeter before, during and after the procedure. The neonate was swaddled, administered 1 mL of oral sucrose, and allowed to suck for 2 minutes prior to the procedure.
- Case (usual measures to control pain plus inhaled lavender essential oil) (Experimental): The neonate was taken to the neonatal unit and monitored with a pulse-oximeter before, during and after the procedure. The neonate was swaddled, administered 1 mL of oral sucrose, and allowed to suck for 2 minutes prior to the procedure. The neonate also had a 7 x 7 cm gauze pad with 1 drop (43.75 mg) of 100% pure LEO (Pranarôm España S.L.) placed 2 cm under their nose for 2 minutes prior to starting the frenotomy and for the duration of the procedure.
  Interventions: Dietary Supplement: Lavender essential oil

INTERVENTIONS:
Dietary Supplement: Lavender essential oil — Use of inhaled lavender essential oil
  Arms: Case (usual measures to control pain plus inhaled lavender essential oil)

SUMMARY:
Clipping of the tongue-tie is a common procedure that neonatologists perform in our neonatal unit to help establish breastfeeding. It is a painful technique where the measures healthcare providers usually perform to control pain (such as sucking) cannot be done at the time of the clipping because the technique is performed on the tongue. The aim of this study was to prove that inhaled lavender essential oil during the clipping of the tongue-tie can help control pain. Participants were newborns born at our hospital during the study period. They were offered to participate and enrolled in the study if their parents agreed to and signed an informed consent. The use of inhaled lavender essential oil is safe. No side effects have been found with its use. The procedure of the frenotomy did not change for patients who were enrolled in the study. By demonstrating that inhaled lavender essential oil helps reduce pain, its use was included as part of the regular measures to control pain during frenotomies at our neonatal unit (Hospital del Mar, Barcelona, Spain). The study started in August 2020 and ended in April 2021.

DETAILED DESCRIPTION:
This randomized clinical trial was conducted with the neonates born at our hospital or less than 15 days old who underwent a frenotomy for type 3 tongue-ties according to Coryllos classification and the Hazelbaker tool during the study period (August 2020 to April 2021). Healthcare providers assessed pain by means of crying time and the highest Neonatal Infant Pain Scale (NIPS) score in the five minutes post procedure, and whether there was an increase in heart rate (HR) and decrease in oxygen saturation (satO2). NIPS evaluates facial expression, crying, breathing pattern, arm and leg position, and state of arousal on a scale from 0 to 7, where 0-2 means no pain to mild pain, 3-4 mild to moderate pain, and >4 severe pain. In an exploratory preliminary study prior to the intervention, a mean (SD) crying time of 19.80 (21.14) seconds was observed. In order to detect a difference of 10 seconds in crying time, a sample size of 71 patients per group was required in order to draw conclusions with a CI 95% and a power of 80%. Patients were enrolled if their parents agreed to and signed a written informed consent.

Data were recorded on demographic (gender, gestational age, birth weight, age in hours at the time of frenotomy) and clinical variables (HR and satO2 before, during, and after the procedure, whether there was crying or not during the procedure, length of crying time in seconds, presence of side effects during the procedure (apnea, desaturation, others) and highest NIPS score within the first 5 minutes after the procedure). The independent variable was the use or not of aromatherapy during frenotomy. The dependent variables were: HR and satO2 pre and post procedure, presence of crying and duration, hours of life at the time of the frenotomy, and the NIPS score. The controlled variables were gestational age, sex, and birth weight.

All the newborns are assessed for the presence of ankyloglossia as part of the routine neonatal evaluation and a frenotomy is offered to all tongue-tied patients. The examiner grades the ankyloglossia based on Coryllos's criteria and the Hazelbaker tool to assess its impact on tongue movement and on breastfeeding. A lingual frenulum is symptomatic if it scores 8 points or less in appearance and/or 11 points or less in function according to Hazelbaker. Advice and help with positioning and attachment for breastfeeding is provided to all the mothers by IBCLC (International Board Certified Lactation Consultant) nurses. During the study period, if a patient with a type 3 tongue-tie was identified, the patient's parents were offered to participate in this study. Accepted patients were allocated into case or control group by simple random sampling using the program OxMAR (Online Minimization and Randomization for Clinical Trials). During the frenotomy the neonate was taken to the neonatal unit and monitored with a pulse-oximeter (COVIDIEN Nellcor Portable SpO2 Patient Monitoring System PM10N, Covidien Ireland Limited, IDA Business & Technology Park, Tullamore, Ireland) before, during and after the procedure. For both groups, neonates were swaddled, administered 1 mL of oral sucrose, and allowed to suck for 2 minutes prior to the procedure. The experimental group also had a 7 x 7 cm gauze pad with 1 drop (43.75 mg) of 100% pure LEO (Pranarôm España S.L.) placed 2 cm under their nose for 2 minutes prior to starting the frenotomy and for the duration of the procedure. The bottle of LEO has a dropper that always dispenses the same amount of oil per drop. The procedure did not start the procedure until the patients were calm and had a NIPS score of 0. Frenotomy was performed by one of the three staff neonatologists using Coryllos' technique: placing a sterile groove director under the tongue straddling the frenulum, holding the frenulum in place with visualization of tongue base and frenulum, and snipping the frenulum with a scissor along the underside of the tongue to its base just proximal to the genioglossus muscle, until a full release is achieved. Once the procedure was completed, the gauze pad was removed and vital signs, whether the baby cried or not, the seconds crying lasted, and the post procedure NIPS score were registered on a data collection sheet. If a neonate cried, calming techniques such as holding, swaddling, and sucking were employed. Following the frenotomy, the neonate was returned to the mother for breastfeeding.

Statistical analysis: Quantitative variables (gestational age, birth weight, age at frenotomy, heart rate pre and post-procedure, increase in heart rate post-procedure, oxygen saturation pre and post-procedure, decrease in oxygen saturation post-procedure, and duration of crying) are described using the mean, standard deviation, and 95% confidence interval (CI); case vs control groups were compared with a Student's t test. Gender, the presence of crying, and adverse effects between the two groups are presented in percentages and compared using Fisher's exact test. NIPS scores between cases and controls were compared with the Wilcoxon rank-sum (Mann-Whitney) test. Statistical significance was set for a p <0.05. Statistical analyses were performed using STATA version 15.1 (StataCorp, College Station, TX, USA).

Our hospital Ethics Committee (CEIm-PSMAR) approved this study (reference code: 2020/9373/I). Prior to patient enrollment, a signed informed consent was obtained from the neonate's parents. This study was conducted according to the ethics code of the Barcelona Medical Association and the principles of the Helsinki-Fortaleza Declaration 2013.

ELIGIBILITY:
Inclusion Criteria:

* Healthy full-term neonates born at Hospital del Mar (Barcelona, Spain), or less than 15 days old who had been discharged and returned for the frenotomy, who underwent a frenotomy for type 3 tongue-ties according to Coryllos classification and the Hazelbaker tool during the study period (August 2020 to April 2021)

Exclusion Criteria:

* Refusal of the patient's parents to participate

Ages: 1 Day to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Crying length | Up to 5 minutes post-procedure
  Crying length after the frenotomy in seconds
NIPS score | Up to 5 minutes post-procedure
  Neonatal Infant Pain Score value (0-7). NIPS evaluates facial expression, crying, breathing pattern, arm and leg position, and state of arousal on a scale from 0 to 7, where 0-2 means no pain to mild pain, 3-4 mild to moderate pain, and >4 severe pain.
Change in heart rate | Up to 5 minutes post-procedure
  Change in heart rate pre/post-procedure (beats per minute)
Change in oxygen saturation | Up to 5 minutes post-procedure
  Change in oxygen saturation (%)

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Fàbregas-Mitjans, Ph.D., Principal Investigator — Hospital del Mar
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fitri SYR, Wardhani V, Rakhmawati W, Pahria T, Hendrawati S. Culturally Based Practice in Neonatal Procedural Pain Management: A Mini Review. Front Pediatr. 2020 Sep 3;8:540. doi: 10.3389/fped.2020.00540. eCollection 2020. PMID 33014934
- [Background] Mitchell A, Boss BJ. Adverse effects of pain on the nervous systems of newborns and young children: a review of the literature. J Neurosci Nurs. 2002 Oct;34(5):228-36. doi: 10.1097/01376517-200210000-00002. PMID 12391738
- [Background] Stevens B, Yamada J, Ohlsson A, Haliburton S, Shorkey A. Sucrose for analgesia in newborn infants undergoing painful procedures. Cochrane Database Syst Rev. 2016 Jul 16;7(7):CD001069. doi: 10.1002/14651858.CD001069.pub5. PMID 27420164
- [Background] Harrison D, Larocque C, Bueno M, Stokes Y, Turner L, Hutton B, Stevens B. Sweet Solutions to Reduce Procedural Pain in Neonates: A Meta-analysis. Pediatrics. 2017 Jan;139(1):e20160955. doi: 10.1542/peds.2016-0955. Epub 2016 Dec 16. PMID 27986905
- [Background] Leng HY, Zheng XL, Yan L, Zhang XH, He HY, Xiang M. [Effects of different types and concentration of oral sweet solution on reducing neonatal pain during heel lance procedures]. Zhonghua Er Ke Za Zhi. 2013 Sep;51(9):654-8. Chinese. PMID 24330983
- [Background] Jones JE, Kassity N. Varieties of alternative experience: complementary care in the neonatal intensive care unit. Clin Obstet Gynecol. 2001 Dec;44(4):750-68. doi: 10.1097/00003081-200112000-00012. No abstract available. PMID 11600855
- [Background] Maya-Enero S, Perez-Perez M, Ruiz-Guzman L, Duran-Jorda X, Lopez-Vilchez MA. Prevalence of neonatal ankyloglossia in a tertiary care hospital in Spain: a transversal cross-sectional study. Eur J Pediatr. 2021 Mar;180(3):751-757. doi: 10.1007/s00431-020-03781-7. Epub 2020 Aug 15. PMID 32803423
- [Background] Lawrence J, Alcock D, McGrath P, Kay J, MacMurray SB, Dulberg C. The development of a tool to assess neonatal pain. Neonatal Netw. 1993 Sep;12(6):59-66. PMID 8413140
- [Background] Lopez V, Nielsen B, Solas M, Ramirez MJ, Jager AK. Exploring Pharmacological Mechanisms of Lavender (Lavandula angustifolia) Essential Oil on Central Nervous System Targets. Front Pharmacol. 2017 May 19;8:280. doi: 10.3389/fphar.2017.00280. eCollection 2017. PMID 28579958
- [Background] Habanananda T. Non-pharmacological pain relief in labour. J Med Assoc Thai. 2004 Oct;87 Suppl 3:S194-202. PMID 21213523
- [Background] Goubet N, Rattaz C, Pierrat V, Bullinger A, Lequien P. Olfactory experience mediates response to pain in preterm newborns. Dev Psychobiol. 2003 Mar;42(2):171-80. doi: 10.1002/dev.10085. PMID 12555281
- [Background] Sadathosseini AS, Negarandeh R, Movahedi Z. The effect of a familiar scent on the behavioral and physiological pain responses in neonates. Pain Manag Nurs. 2013 Dec;14(4):e196-e203. doi: 10.1016/j.pmn.2011.10.003. Epub 2012 Feb 28. PMID 24315273
- [Background] Mikami-Saito Y, Maekawa M, Wada Y, Kanno T, Kurihara A, Sato Y, Yamamoto T, Arai-Ichinoi N, Kure S. Essential oils can cause false-positive results of medium-chain acyl-CoA dehydrogenase deficiency. Mol Genet Metab Rep. 2020 Nov 5;25:100674. doi: 10.1016/j.ymgmr.2020.100674. eCollection 2020 Dec. PMID 33204637
- [Result] Goubet N, Strasbaugh K, Chesney J. Familiarity breeds content? Soothing effect of a familiar odor on full-term newborns. J Dev Behav Pediatr. 2007 Jun;28(3):189-94. doi: 10.1097/dbp.0b013e31802d0b8d. PMID 17565285
- [Result] Johnston CC, Fernandes AM, Campbell-Yeo M. Pain in neonates is different. Pain. 2011 Mar;152(3 Suppl):S65-S73. doi: 10.1016/j.pain.2010.10.008. Epub 2010 Oct 23. PMID 20971562
- [Result] Razaghi N, Aemmi SZ, Sadat Hoseini AS, Boskabadi H, Mohebbi T, Ramezani M. The effectiveness of familiar olfactory stimulation with lavender scent and glucose on the pain of blood sampling in term neonates: A randomized controlled clinical trial. Complement Ther Med. 2020 Mar;49:102289. doi: 10.1016/j.ctim.2019.102289. Epub 2019 Dec 26. PMID 32147068
- [Result] Akcan E, Polat S. Comparative Effect of the Smells of Amniotic Fluid, Breast Milk, and Lavender on Newborns' Pain During Heel Lance. Breastfeed Med. 2016 Aug;11(6):309-314. doi: 10.1089/bfm.2015.0174. Epub 2016 Jun 17. PMID 27315487
- [Result] Vaziri F, Khosropoor M, Hidari M, Pourahmad S, Morshed Behbahani B, Saki F. The Effect of Aromatherapy by Lavender Oil on Infant Vaccination Pain: a Double Blind Randomized Controlled Trial. J Caring Sci. 2019 Mar 1;8(1):17-21. doi: 10.15171/jcs.2019.003. eCollection 2019 Mar. PMID 30915309
- [Result] Cetinkaya B, Basbakkal Z. The effectiveness of aromatherapy massage using lavender oil as a treatment for infantile colic. Int J Nurs Pract. 2012 Apr;18(2):164-9. doi: 10.1111/j.1440-172X.2012.02015.x. PMID 22435980
- [Result] Field T, Field T, Cullen C, Largie S, Diego M, Schanberg S, Kuhn C. Lavender bath oil reduces stress and crying and enhances sleep in very young infants. Early Hum Dev. 2008 Jun;84(6):399-401. doi: 10.1016/j.earlhumdev.2007.10.008. Epub 2007 Nov 28. PMID 18053656